CLINICAL TRIAL: NCT05827029
Title: Comparison of Gastric Residual Volume After Ingestion of Carbohydrate Drink and Water in Obese Volunteers: A Randomized Crossover Study
Brief Title: Gastric Volume After Ingestion of Carbohydrate Drink vs Water in Obese Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Chanatthee Kitsiripant, Asst.Prof., Prince of Songkla University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Screening
Other Study IDs: REC.65-236-8-1
Record Dates: First submitted 2023-04-09; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Obesity; Gastric Emptying
Keywords: gastric residual volume, obesity, carbohydrate drink
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative carbohydrate drink (Experimental)
  Interventions: Procedure: Preopertive drink
- Water (Placebo Comparator)
  Interventions: Procedure: Preopertive drink

INTERVENTIONS:
Procedure: Preopertive drink — * Group C: will receive a carbohydrate drink of 400 ml (50 g of glucose prepared by nutrition division, same appearance and containing bottles of water)
  * Group W: will receive water 400 ml (prepared by nutrition division, Songklanagarind hospital, same appearance and containing bottles of carbohydrate drink) In both groups, the received 400-mL drink was consumed within 5 minutes.
  * Before drinking, baseline data (gastric residual volume, POCT glucose, degree of hunger, and thirst) will be evaluated.
  * Gastric ultrasound will be performed by the same Radiologist on each participant at 0, 30, 60, 90, 120 minutes
  * after drinking to evaluate the gastric residual volume and time to empty gastric antrum.
  * POCT glucose and degree of hunger and thirst are also assessed again at 120 minutes after drinking.
  * After completing one type of drinking, participants will be appointed again after 1 week later for doing the same protocol with another drinking.

SUMMARY:
This randomized crossover study compares gastric residual volume after ingestion of carbohydrate drinks and water in obese volunteers. The main question[s] it aims to answer are:

* Is it safe for obese patients to shorten their fasting by allowing preoperative drinks?
* How long is the gastric emptying time in obese patients? Participants also will be evaluated the level of thirst/hungry and blood sugar.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age 18 - 65 years old
* BMI ≥ 30 kg/m2
* NPO for at least 6 hours before the study

Exclusion Criteria:

* Diabetes Mellitus
* Chronic kidney disease or End-stage renal disease
* Use of any medication that affects gastric secretion or emptying (Histamine 2 receptor antagonist eg. Ranitidine/Proton pump inhibitor eg. Omeprazole/Acid neutralization eg. Aluminium hydroxide/Prokinetic eg. Domperidone) within the past 24 hours
* Gastroesophageal reflux disease
* Pregnancy
* History of upper gastrointestinal surgery
* In diet program or use appetite suppressant drug (eg. Liraglutide, Naltrexone, Phentermine, Diethylpropion) within the past 24 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
gastric residual volume | baseline and every 30 minutes until 2 hours after drinking
  changes in gastric residual volume during 2 hours after drinking

SECONDARY OUTCOMES:
time to empty gastric antrum | baseline and 120 minutes after drinking
POCT glucose | baseline and 120 minutes after drinking
  changes in glucose level after ingest carbohydrate drink or water
thirst and hunger level | baseline and 120 minutes after drinking
  thirst and hunger level will be evaluated by visual rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Chanatthee Kitsiripant, Principal Investigator — Department of Anesthesiology, Faculty of Medicine, Prince of Songkla University
Locations (1):
- Department of Anesthesiology, Faculty pf Medicine, Songkhla, Thailand